CLINICAL TRIAL: NCT02387489
Title: A Randomized Clinical Trial of Screening, Brief Intervention, and Referral-to-Treatment (SBIRT) Services in School-based Health Centers
Brief Title: A Clinical Trial of SBIRT Services in School-based Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-03-221; 1R01DA036604 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-13 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Marijuana Use; Alcohol Consumption; Unsafe Sex; Risk Behavior
MeSH Terms: conditions — Marijuana Use; Alcohol Drinking; Unsafe Sex; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBI (Active Comparator): Nurse-delivered Brief Intervention
  Interventions: Behavioral: Brief in-person motivational intervention
- CBI (Experimental): Computerized Brief Intervention
  Interventions: Behavioral: Computerized Brief Intervention

INTERVENTIONS:
Behavioral: Brief in-person motivational intervention — Brief in-person motivational intervention tailored to participants' risk behaviors, delivered by a nurse.
  Arms: NBI
Behavioral: Computerized Brief Intervention — Computer-delivered motivational intervention tailored to participants' risk behaviors.
  Arms: CBI

SUMMARY:
The purpose of the study is to examine the comparative effectiveness of a computerized brief intervention vs. an in-person brief intervention delivered by a nurse in reducing marijuana, alcohol, and sex risk behaviors in adolescents receiving services in school-based health centers.

DETAILED DESCRIPTION:
Substance use among adolescents continues to be highly prevalent in the US. Likewise, many adolescents engage in sexual behaviors that place them at elevated risk for HIV and other sexually transmitted infections. Screening, brief intervention, and referral to treatment (SBIRT) is a promising approach for integrating substance use services into healthcare settings. School-based health centers (SBHCs) are a rapidly expanding model of healthcare delivery offering health services far beyond those of the traditional school health office. Implementing SBIRT in SBHCs could have major public health benefits, but research is needed to identify the most effective way to deliver SBIRT for adolescents in these settings. Two approaches for SBIRT that are particularly promising in their practicality, scalability, and sustainability are nurse practitioner-delivered brief intervention and computer-delivered brief intervention. This randomized controlled trial seeks to determine the comparative clinical effectiveness and cost-effectiveness of these two approaches in reducing marijuana use, alcohol use, and sex risk behaviors. The study will be conducted in SBHCs embedded within public high schools in Baltimore, Maryland. SBHC patients will be screened for eligibility by research staff with the CRAFFT, a brief substance misuse screening instrument recommended by the American Academy of Pediatrics. The study will enroll 300 male and female adolescents who report risky marijuana or alcohol use. Participants will be randomly assigned to receive a nurse practitioner-delivered brief intervention (NBI) consisting of brief motivational advice as part of their medical visit, or a promising interactive computer-delivered brief intervention (CBI) based on motivational interviewing. Both intervention conditions will include HIV risk reduction content tailored based on individual risk factors, and both conditions will include a referral pathway for additional substance abuse assessment and possible treatment by specialized substance abuse treatment staff. Research assessments will be conducted at baseline and at 3- and 6-month follow-up, and will gather self-reported data on substance use and sexual risk behaviors. A focused economic analysis will compare the NBI and CBI conditions with respect to their incremental cost-effectiveness for selected primary behavioral outcomes and for quality-adjusted life years (QALYs). A qualitative process evaluation will examine adolescent participants' and SBHC staff members' perspectives on the competing BI strategies. This study has the potential for significant public health impact because it could identify the most effective SBIRT model for addressing adolescent substance use and HIV risk behaviors, both of which can have major health repercussions in the near-term and over the lifespan. The study is highly innovative in its focus on SBHCs, a rapidly expanding healthcare model that is uniquely suited to maximize the impact and reach of SBIRT for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen at one of the participating school-based health centers
* Self-reported marijuana or alcohol use (on CRAFFT screener)
* CRAFFT score of 2 or higher

Exclusion Criteria:

* use of illicit drugs, or non-medical use of prescription drugs, other than marijuana, alcohol, or tobacco (as self-reported on CRAFFT screener)
* current enrollment in substance abuse treatment
* pregnancy

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
frequency of marijuana use | 3 months; 6 months
  days of marijuana use in the past 30 days

SECONDARY OUTCOMES:
frequency of alcohol use | 3 months; 6 months
  days of alcohol use in the past 30 days
binge drinking | 3 months; 6 months
  binge drinking in the past 30 days
Marijuana Risks | 3 months; 6 months
  Marijuana ASSIST risk scores
Alcohol Risks | 3 months; 6 months
  Alcohol ASSIST risk scores
Unprotected sex | 3 months; 6 months
  Days of unprotected sex
Sex while intoxicated | 3 months; 6 months
  Days of sex while under the influence of drugs or alcohol

OTHER OUTCOMES:
Assessment/treatment entry | 3 months; 6 months
  access assessment or treatment services